CLINICAL TRIAL: NCT03114111
Title: Pilot Study for the Use of Photodynamic Therapy in the Treatment of Seborrheic Dermatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 408732
Record Dates: First submitted 2017-02-14; First posted 2017-04-14 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Application of ALA (Active Comparator): The treatment will consist of split-face comparisons of no application of aminolevulinic acid (ALA) vs ALA application to either half of the face. Prior to ALA application, the face will be swabbed for microbiome analysis. After the ALA application, the subjects will incubate with the ALA on their face per the standard PDT protocol used at UC Davis Dermatology clinic for facial PDT treatments. The side of the face being treated will remain the same during all treatments.
  Interventions: Drug: aminolevulinic acid (ALA)
- No Application of ALA (Placebo Comparator): For the placebo, Demo Levulan Kerastick, which contains no active ingredient and is enclosed in same cardboard sleeve and cap, will be applied to the other side of the face to mimic the surface of the ALA application stick. After the placebo application, the subjects will incubate with the placebo on their face per the standard PDT protocol used at UC Davis Dermatology clinic for facial PDT treatments. The side of the face being treated will remain the same during all treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aminolevulinic acid (ALA)
  Other Names: LEVULAN® KERASTICK®
  Arms: Application of ALA
Drug: Placebo
  Other Names: Demo Levulan Kerastick
  Arms: No Application of ALA

SUMMARY:
The purpose of this study is:

1. To determine the efficacy of photodynamic therapy (PDT) in the treatment of seborrheic dermatitis.
2. To determine how PDT alters the skin microbiome in subjects with seborrheic dermatitis before and after treatment.
3. To determine how PDT alters sebum secretion rates in subjects with seborrheic dermatitis before and after treatment.

The researchers hypothesize that PDT will be efficacious in the treatment of seborrheic dermatitis.

DETAILED DESCRIPTION:
This pilot project investigates the use of PDT may be useful in the treatment of seborrheic dermatitis based on the following: The Malassezia spp is capable of forming biofilms, 2) PDT has been shown to be effective against Malassezia spp PDT can break up bioflims of both bacterial and fungal origin and benzoyl peroxide, a prooxidant treatment similar to PDT, has been shown to be effective in the treatment of seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects 18 years or older with seborrheic dermatitis of the face will be included.

Exclusion Criteria:

* Subjects who are taking systemic corticosteroids (at doses of prednisone greater than or equal to 5 mg daily), antibiotics (PO, IM or IV) or using topical anti- fungals, steroids, antibiotics, permethrin, or calcineurin inhibitors within 2 weeks prior to the study will be excluded.
* The exclusion criteria will also include the presence of other untreated inflammatory conditions (such as lupus, atopic dermatitis, or psoriasis) or untreated malignancies on the face (including skin cancers such as basal cell carcinoma, squamous cell carcinoma and melanoma).
* Any subjects with known or suspected hypersensitivity to any constituent of the study medication or a history of photosensitivity due to conditions such as lupus erythematosus and porphyria will be excluded.
* Subjects who have had photodynamic therapy (PDT) to the face for any reason within the past year will be excluded as well.
* Adults unable to consent, individuals under the age of 18, pregnant or breastfeeding women and prisoners will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
severity of seborrheic dermatitis before and after ALA treatment as determined by Seborrhea Area and Severity Index Face (SASI-F) | up to 3 months

SECONDARY OUTCOMES:
microbiome analysis before and after ALA treatment | up to 3 months
facial sebum production rates before and after ALA treatment | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT03114111/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03114111/ICF_001.pdf